CLINICAL TRIAL: NCT00268723
Title: An Efficacy Study of Single-Dose Levalbuterol Tartrate HFA MDI Versus Placebo in Prevention of EIB in Subjects 18 Years of Age and Older With EIB
Brief Title: Efficacy Study of Single-Dose Levalbuterol Tartrate HFA MDI Vs Placebo in Subjects 18 Years and Older With EIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 051-925
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Exercise-induced Bronchospasm
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): levalbuterol HFA MDI 90 mcg QID
  Interventions: Drug: Levalbuterol tartrate HFA MDI
- 2 (Placebo Comparator): Placebo MDI QID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levalbuterol tartrate HFA MDI — levalbuterol MDI 90 mcg QID
  Other Names: Xopenex MDI
  Arms: 1
Drug: Placebo — Placebo MDI QID
  Arms: 2

SUMMARY:
To determine if administration of levalbuterol tartrate HFA MDI in subjects with EIB will be effective in the prevention of EIB and be safe and well-tolerated.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, multicenter, two-way crossover study of levalbuterol tartrate HFA MDI in subjects 18 years of age and older with EIB. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Subjects were males or females and 18 years of age or older at the time of consent.
* Female subjects considered not of childbearing potential were either surgically sterile or greater than one-year postmenopausal, defined as a complete cessation of menstruation for at least one year.
* Female subjects of child-bearing potential had a negative urine pregnancy test at screening.
* Female subjects of child-bearing potential agreed to use an acceptable method of birth control throughout the study.
* Subjects were in good health and were not suffering from any chronic condition that might affect their respiratory or cardiac function (including cardiac arrhythmias).
* Subjects had a documented diagnosis of exercise-induced bronchospasm for a minimum of 6 months prior to study start.
* Subjects had stable baseline asthma and had been using a beta2-adrenergic agonist, and/or anti-asthma anti-inflammatory medication, and/or over-the-counter asthma medication for at least 6 months prior to study start.

Exclusion Criteria

* Subjects with currently diagnosed life-threatening asthma defined as a history of: asthma episodes requiring intubation, associated hypercapnia, respiratory arrest, or hypoxic seizures within 12 months prior to study start.
* Subjects with a history of hospitalization for asthma within 4 weeks prior to study start, or who were scheduled for in-patient hospitalization, including elective surgery, during the course of the trial.
* Subjects with a documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis.
* Subjects who suffered from a clinically significant upper or lower respiratory tract infection in the 3 weeks prior to study start.
* Subjects with any clinically significant unstable medical abnormality, chronic disease (other than asthma), or history of a clinically significant abnormality of the cardiovascular, gastrointestinal, respiratory, hepatic, renal, endocrine, or central nervous systems that was not currently well controlled by medication or that may have interfered with the successful completion of the protocol.
* Subjects with a history of cancer (exception: basal-cell carcinoma in remission for a minimum of 5 years).
* Subjects with a known sensitivity to levalbuterol, racemic albuterol, or any of the excipients contained in any of these formulations.
* Subjects using any prescription drug with which levalbuterol tartrate administration is contraindicated.
* Subjects with a history of substance abuse or drug abuse within 12 months preceding study start.
* Subjects who participated in an investigational drug study within 30 days prior to study start, or who were currently participating in another clinical trial.
* Subjects with a greater than 10-pack-year history of cigarette smoking or use of any tobacco products within 6 months of study start.
* Subject was a staff member or relative of a staff member.
* Subjects with unstable asthma, or had a change in asthma therapy, or a visit to the emergency department or hospital for worsening asthma within 4 weeks of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-12; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
maximum percent FEV1 decrease from visit postdose/prechallenge | Days 1, 4, 7

SECONDARY OUTCOMES:
FEV1 area under the curve (AUC0-60 mins) (% decrease from visit postdose/prechallenge) | Days 1, 4, 7
time to FEV1 recovery | Days 1, 4, 7
minimum percent change in FEV1 from visit postdose/prechallenge | Days 1, 4, 7
minimum percent change in FEV1 from visit predose | Days 1, 4, 7
protected/unprotected subject counts (unprotected: >20% decrease; moderately protected: 10% to 20% decrease; and protected: <10% decrease from postdose/prechallenge FEV1) | Days 1, 4, 7
percent change in FEV1 from predose to postdose/prechallenge | Days 1, 4, 7

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Denver, Colorado
  - Burke, Virginia